CLINICAL TRIAL: NCT00841412
Title: Prevention of Weight Loss in Long-Term Care Veterans
Brief Title: Prevention of Weight Loss in Long Term Care Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIR 07-250
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-10

CONDITIONS: Malnutrition
Keywords: Usual Care Control Group
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Intervention Group (Experimental): Immediate Intervention: Long term care units assigned to the Immediate Intervention group were first to receive the staff training and management intervention to improve nutritional care processes.
  Interventions: Behavioral: Immediate Intervention Group
- Delayed Intervention Group (Active Comparator): Delayed Intervention: Long term care units assigned to the Delayed Intervention group were monitored under usual care conditions to serve as a control for the Immediate Intervention group. Then, these units received the staff training and management intervention at a later date.
  Interventions: Behavioral: Delayed Intervention Group

INTERVENTIONS:
Behavioral: Immediate Intervention Group — Unit staff received weekly training and feedback for 12-weeks to improve daily nutritional care processes.
  Arms: Immediate Intervention Group
Behavioral: Delayed Intervention Group — Research staff monitored this group under usual care conditions, then these units crossed over into intervention.
  Arms: Delayed Intervention Group

SUMMARY:
Background: Numerous studies have shown that many LTC residents receive inadequate staff assistance with eating, which places them at risk for under-nutrition, dehydration and weight loss. Moreover, improvements in feeding assistance care have been shown to improve residents' daily food and fluid consumption and weight loss outcomes.

Objectives: The purpose of this program evaluation project is to train indigenous LTC staff how to improve nutritional care within the constraints of existing staffing resources.

Methods: A multiple baseline design was used to evaluate the effectiveness of the program in one federal and one state VA LTC facility. Research staff collected baseline measures related to nutritional care processes and resident outcomes. All LTC units in each of the two sites were divided into two groups for program implementation. The program was implemented with staff and residents on the units in the immediate intervention group; while, the delayed intervention group remained in usual care and continued to be monitored monthly for all care process and resident outcome measures.

Status: This project ended 10/1/13. Five published papers resulted from this study.

DETAILED DESCRIPTION:
Background:

Numerous studies have shown that many long term care (LTC) residents receive inadequate staff assistance with eating, which places them at risk for under-nutrition, dehydration and weight loss. Moreover, improvements in feeding assistance care have been shown to improve residents' daily food and fluid consumption and weight loss outcomes. However, these improvements have only been achieved through the use of research staff as opposed to indigenous LTC staff due to staffing resource limitations that exist in most LTC facilities. The purpose of this program evaluation project is to train indigenous LTC staff how to improve nutritional care within the constraints of existing staffing resources.

Objectives:

The PI of this proposal has developed standardized assessment, monitoring and staffing needs projection tools that can be used by long-term care (LTC) providers to improve feeding assistance care delivery and unintentional weight loss outcomes. The primary objective of this project is to train indigenous LTC staff how to (1) identify residents in need of feeding assistance, (2) effectively monitor daily care delivery; and, (3) utilize existing, non-nursing staff for some mealtime tasks to improve care.

Methods:

A multiple baseline design was used to evaluate the effectiveness of the program in one federal and one state VA long-term care (LTC) facility. Research staff collected baseline measures related to organizational characteristics, including staffing, nutritional care processes and resident outcomes including oral food and fluid intake and weight status. All LTC units in each of the two sites were divided into two groups for program implementation purposes (for a total of 4 groups across the 2 sites) based on the proximity of a unit to other units, resident and staff characteristics. The program was implemented with staff and residents on the units in the first site/group; while, the second site/group remained in usual care and continued to be monitored monthly for all care process and resident outcome measures. Research staff trained LTC staff in the implementation of program protocols during a 12-week intervention period. Research staff then monitored LTC staff implementation of the program monthly following intervention to determine the sustainability of the program in the absence of research staff. All staff training and monitoring was repeated for the LTC units in groups three and four. The intent of this program evaluation study was to determine the effectiveness and cost of translating efficacious research protocols into care practice to improve the nutritional status of LTC veterans.

Status: This study is officially complete.

ELIGIBILITY:
Inclusion Criteria:

* Long-stay,
* free of feeding tube,
* not receiving hospice care,
* not on a planned weight loss diet,
* able to speak English

Exclusion Criteria:

* short stay/rehab only
* feeding tube
* hospice
* planned weight loss diet

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 222 (Actual)
Dates: Start 2009-02; Primary Completion 2011-10 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra F Simmons, BA MA PhD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

REFERENCES:
- [Result] Simmons SF, Durkin DW, Shotwell MS, Erwin S, Schnelle JF. A staff training and management intervention in VA long-term care: impact on feeding assistance care quality. Transl Behav Med. 2013 Jun;3(2):189-99. doi: 10.1007/s13142-013-0194-3. PMID 24073169
- [Result] Simmons SF, Sims N, Durkin DW, Shotwell MS, Erwin S, Schnelle JF. The quality of feeding assistance care practices for long-term care veterans: implications for quality improvement efforts. J Appl Gerontol. 2013 Sep;32(6):669-86. doi: 10.1177/0733464811433487. Epub 2012 Mar 22. PMID 25474793
- [Result] Durkin DW, Shotwell MS, Simmons SF. The impact of family visitation on feeding assistance quality in nursing homes. J Appl Gerontol. 2014 Aug;33(5):586-602. doi: 10.1177/0733464814522126. Epub 2014 Feb 18. PMID 24652932
- [Result] Durkin DW, Umayam SP, Sims N, Cleeton P, Simmons SF. Whom do veteran nursing home residents prefer to talk to about satisfaction with care?: implications for nursing staff. J Gerontol Nurs. 2012 Dec;38(12):38-45. doi: 10.3928/00989134-20121109-01. PMID 23189996
- [Result] Simmons SF, Durkin DW, Rahman AN, Schnelle JF, Beuscher LM. The value of resident choice during daily care: do staff and families differ? J Appl Gerontol. 2014 Sep;33(6):655-71. doi: 10.1177/0733464812454010. Epub 2012 Aug 1. PMID 25143465

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Intervention Group/Units: Immediate Intervention units received a staff training and management intervention to improve daily nutritional care processes.
- Delayed Intervention Group/Units: Delayed Intervention units (control group) was monitored by research staff under usual care conditions.
Period: Overall Study
Arm/Group | Immediate Intervention Group/Units | Delayed Intervention Group/Units
Started | 120 (200 of 222 consented residents completed baseline assessments across both groups.) | 80 (80 residents were in the delayed intervention group, but all residents received intervention.)
Completed | 80 (130 residents completed all study phases across both groups, including follow-up.) | 50
Not Completed | 40 | 30

BASELINE CHARACTERISTICS:
Population: 200 long-stay veterans completed baseline assessments.
Groups:
- Overall (Both Groups Combined): Participants were randomized by unit and each unit received intervention so characteristics of participants are reported overall for both groups combined.
Arm/Group | Overall (Both Groups Combined)
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.00 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 171
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 200

OUTCOME MEASURES:

1. Primary Outcome: Quality of Feeding Assistance Care Processes
Description: Research staff observed each participant during six meals per study phase. Research staff documented the total amount of staff time spent providing feeding assistance and each type of assistance per resident per meal. These data were used to construct standardized "feeding assistance care quality indicators" wherein the number of resident meal observations was variable. For example, one indicator was defined as: Percentage of meals during which resident intake was below 50% and staff offered and alternative to the served meal". Thus, the denominator for total number of observed meals scored varied by indicator. There were multiple indicators; thus, there is inadequate space to provide an adequate description of each measure and the corresponding scoring rules here. Please refer to published papers for a complete description of all outcome measures.
Time Frame: 3 month intervention and 3 month follow up periods
Population: Each participants was observed during six scheduled meals per person per study phase. A total of 130 participants completed all study phases and had complete data for analyses.
Measure: Number; unit: percentage of meal observations
Units Other Than Participants: Meal Observations
Groups:
- Overall (Both Groups Combined): Participants were randomized by unit and each unit received intervention so outcome measures are reported overall for both groups combined.
Arm/Group | Overall (Both Groups Combined)
Number analyzed (Participants) | 130
Number analyzed (Meal Observations) | 1560
percentage of meal observations
  Percent of Meals with Accurate Chart Documentation | 66.7
  Percent of Meals with Social Interaction | 47.2
  Percent of Meals with Assistance | 61.4
Statistical Analysis 1: Comparison: Overall (Both Groups Combined); Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.59 to 0.96] — The above results are for just one of multiple feeding assistance care process measures: proportion of meals during which residents received assistance to eat baseline to post intervention

ADVERSE EVENTS:
Time Frame: Three months of Intervention
Arm/Group | Overall (Both Groups Combined)
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

LIMITATIONS AND CAVEATS:
This study was conducted in only two VA facilities in one geographic region with predominately White, male residents. All study results have been published in a series of papers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes